CLINICAL TRIAL: NCT00645216
Title: A Phase 1, Open Label, Randomized, Fixed Sequence Study To Evaluate The Effect Of Multiple Dose Administration Of Grapefruit Juice On The Multiple Dose Pharmacokinetics Of CP-945,598 In Healthy Overweight And Obese Subjects
Brief Title: Study Examing The Effect of Grapefruit Juice On The Blood And Urine Samples of Study Drug And Its By Product And Safety
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A5351047
Record Dates: First submitted 2008-03-20; First posted 2008-03-27 (Estimated); Last update posted 2009-08-10 (Estimated); Status verified 2008-03

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CP-945,598 with Grapefruit Juice (Experimental): CP-945,598 with Grapefruit Juice
  Interventions: Drug: CP-945,598
- CP-945,598 alone (Experimental): CP-945,598 alone
  Interventions: Drug: CP-945,598

INTERVENTIONS:
Drug: CP-945,598 — Subjects take CP-945,598 alone for 21 days
  Arms: CP-945,598 alone
Drug: CP-945,598 — Subjects take CP-945,598 from Days 1 to 7, then take CP-945,598 and Grapefruit Juice from Days 8 to 21
  Arms: CP-945,598 with Grapefruit Juice

SUMMARY:
CP-945,598 is eliminated primarily by enzyme CYP3A. Grapefruit juice may affect the activity of CYP3A and alter the amount of CP-945,598 in the blood. This study will therefore compare the time course of drug concentrations in the body, safety and tolerability of CP-945,598 given with or without grapefruit juice in healthy obese/overweight subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female subjects between the ages of 18 and 55 years.
2. Body Mass Index (BMI) of 27 to 40 kg/m2.
3. Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other trial procedures.

Exclusion Criteria:

* Non-prescribed use of drugs of abuse/ recreational drugs;
* Recent treatment with experimental drugs or herbal experiments;
* EKG and blood pressure parameters falling outside of protocol-specified limits;
* History of regular alcohol or tobacco use exceeding protocol-specified limits; grapefruit juice intolerance.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2007-06; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Measurement of durg and metabolite concentrations in serum from blood sampling collected at various times over 24 hours dosing interval on Day 7 and 21, before dosing on days 5,6, 12, 13, 14, 19 and 20. | 21 days
Safetey laboratory tests (chemistry, hematology, urinalysis) on Days -1 and 22 | 21 days
Adverse event monitoring throughout duration of the study | 21 days

SECONDARY OUTCOMES:
Urinary 6-β-hydroxycortisol:cortisol ratios (CMR) on Days 0 and 21. | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5351047&StudyName=Study%20Examing%20The%20Effect%20of%20Grapefruit%20Juice%20On%20The%20Blood%20And%20Urine%20Samples%20of%20Study%20Drug%20And%20Its%20By%20Product%20And%20Safety